CLINICAL TRIAL: NCT05118815
Title: Characterization and Behavior of Peri-implant Tissues on the New Anti-rotational Slim Abutment Galimplant. Single-blind Randomized Multicenter Clinical Trial.
Brief Title: Peri-implant Tissues on the Galimplant Anti-rotational Slim Abutment.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: University of Salamanca (Other); University of Valencia (Other); Universidad de Murcia (Other); Health Research Institute of Santiago (Other)
Responsible Party: Principal Investigator, Mario Pérez Sayáns, Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MC/TP/2021
Record Dates: First submitted 2021-10-16; First posted 2021-11-12 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Teeth Absent; Tooth-loss; Tooth Extraction; Dental Implant
Keywords: oral rehabilitation; dental implants; marginal bone loss; periimplant tissues; abutments
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Intervention Model Description: A total of 60 dental implants Hexagonal Internal Connection Implants (Model IPX), Galimplant® will be used in this study, for the replacement of bilateral maxillary posterior missing teeth in 30 patients (split-mouth study). For the designation of the type of transepithelial abutment to be placed in each hemimaxillary, we will use an online randomization service (www.randomization.com). After surgery, 30 patients will have a conventional straight esthetic abutment 3 mm in height (control group), and the other 30 will have a Slim (New Slim) transepithelial abutment of the same height (test group); in no case will we place the transepithelial closure abutment to achieve contact of the peri-implant mucosa with the surface of the transepithelial abutments. The implant will be placed whenever bone and gingival availability allows it juxta-osseous to avoid collateral damage in the exeresis of the peri-implant perimetral soft tissue (hereinafter donut)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional straight esthetic abutment (Active Comparator): After implant surgery, 30 patients will have a 3 mm high conventional straight esthetic abutment placed. The implant placement will follow the manufacturer's instructions and the operator's expertise to achieve stability with an insertion torque of at least 40 N, recording the final torque with a calibrated torque wrench. The implant will be placed whenever bone and gingival availability allows it, juxta-osseous to avoid collateral damage in the peri-implant perimetral soft tissue excision (donut). The abutment will be placed at 30 N as indicated by the manufacturer. After removal of the donut, a new abutment will be placed and left in place up to 3 months to allow healing and complete osseointegration. Patients will receive prosthodontic loading following standard metal-ceramic rehabilitation protocols and the manufacturer's recommendation. The prosthesis will be screw-retained, on the abutment placed after excision of the donut, screwed at 25 N.
  Interventions: Other: Standard abutment
- Slim (New Slim) transepithelial abutment (Experimental): After surgery, 30 patients will have a 3 mm high transepithelial New Slim abutment placed. The implant placement will follow the manufacturer's instructions and the operator's expertise to achieve stability with an insertion torque of at least 40 N, recording the final torque with a calibrated torque wrench. The implant will be placed whenever bone and gingival availability allows it, juxta-osseous to avoid collateral damage in the peri-implant perimetral soft tissue excision (donut). The abutment will be placed at 30 N as indicated by the manufacturer. After removal of the donut, a new abutment will be placed and left in place up to 3 months to allow healing and complete osseointegration. Patients will receive prosthodontic loading following standard metal-ceramic rehabilitation protocols and the manufacturer's recommendation. The prosthesis will be screw-retained, on the abutment placed after excision of the donut, screwed at 25 N
  Interventions: Other: Slim abutment

INTERVENTIONS:
Other: Slim abutment — Use a narrower abutment to see if they present a better biological seal.
  Arms: Slim (New Slim) transepithelial abutment
Other: Standard abutment — Use a standard abutment
  Arms: Conventional straight esthetic abutment

SUMMARY:
A dental implant is an alloplastic material surgically inserted in a residual bone ridge, mainly with a prosthetic foundation. Nowadays the most widely used implants and with a higher degree of scientific evidence are the titanium root-form endosseous implants. In addition to the root component, the prosthodontic systems that allow the crown to be connected to the implant are very important. The aim of this project is to compare a classic anti-rotational straight esthetic multi-position attachment with the new anti-rotational straight esthetic slim multi-position abutment, both placed at the time of implant surgery. A multicenter randomized single-blind (for the patient) split-mouth randomized clinical trial will be performed to compare the composition, distribution and structure of the peri-implant tissues around the classic straight (control) and Slim (test) intermediate prosthetic abutments of the manufacturer Galimplant (Sarria; Lugo, Spain). The objective is to study which abutment design obtains a better biological seal from the clinical and histomorphometric point of view. For this purpose, 60 dental implants will be placed for the replacement of bilateral posterior absences in 30 patients attending the Master of Oral Medicine, Oral Surgery and Implantology of the University of Santiago de Compostela, Spain.

DETAILED DESCRIPTION:
Throughout implantological history there have been many proposals and modifications in terms of anchorage system, shape, materials, etc. In this project we intend to compare a classic anti-rotational straight esthetic multi-position attachment with the new anti-rotational straight esthetic slim multi-position abutment.

This will hypothetically allow to increase the contact surface of the peri-implant connective tissue, increase the adhesion and sealing power, improve the biological width and consequently minimize the risk of peri-implant diseases such as mucositis and peri-implantitis.

In this regard, we must analyze the healing process of the peri-implant soft tissue after surgery, which will result in a stable peri-implant mucosa. After surgery, soft tissue healing around the transmucosal portion of an implant begins with the formation of a blood clot and the induction of an inflammatory process aimed at tissue formation and remodeling. If that soft tissue formation and remodeling is adequate, the healing process will result in an effective attachment mucosa around the transmucosal portion of the implant.

To obtain this adequate peri-implant mucosa, it is very important that a proper healing process takes place. This process includes the recruitment of inflammatory cells and a process of angiogenesis; and if both processes are correctly developed, all the phases of mucosal healing (hemostasis, inflammation, proliferation, and remodeling of the collagen matrix) will occur successfully.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all the inclusion criteria and none of the exclusion criteria will be informed verbally and in writing about the study and will sign the informed consent form provided for their participation.
* Systemic conditions favorable for the performance of oral surgical procedures (ASA I/II).
* Not to be completely edentulous
* Bilateral absence of at least two teeth (one per hemimaxillary) in the posterior area (from the first premolar to the second molar) with or without free distal ends.
* That do not require regenerative techniques
* That allow the placement of Galimplant implants of 4.5 or 5 mm in diameter in edentulous areas with mature bone of at least 3 months healing time
* With a prosthetic space of at least 8 mm.
* In case of odd absences, a slim abutment will be placed, being the group to be tested always in the majority.

Exclusion Criteria:

* Presence of any disease, condition or medication that may compromise the healing and/or osseointegration of dental implants (uncontrolled diabetes mellitus, immunosuppression, administration of bone modifying agents (BMA). Presence of any severe mental disorder, and patients who have received head and neck radiotherapy during the previous 18 months.
* Patients who do not have sufficient peri-implant keratinized gingiva to allow at least 1 mm of residual gingiva after excision of the tissue under study.
* Esthetic edentulous areas of 13-23, Implants with primary stability with ISQ < 50 or <40N, or with abutments that cannot receive torque at 30N are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2025-07-29 (Estimated)

PRIMARY OUTCOMES:
Peri-implant mucosa located around conventional esthetic abutments and the new Slim Galimplant abutments | 3 months
  To histologically and immunohistochemically compare the peri-implant mucosa through a sample of peri-implant mucosa by means of a section around the transepithelial abutment, obtaining a 1.5-2 mm sample that will be fixed in 10% formaldehyde and transferred to the University of Murcia for histological and immunohistochemical study. The portion of peri-implant mucosa will be deparaffinised and two sections of 5 µm each will be obtained. One, stained with HE and analysed with software Image J version 1.46, calculating the average of 25 thickness measurements for each of the samples.The other 5 µm section will be stained with Masson-Goldner trichrome as a birefringent stain to facilitate the accuracy of the study.

SECONDARY OUTCOMES:
Inflammatory response rate | 3 months
  To compare the inflammatory response of the peri-implant mucosa located around conventional esthetic abutments and the new Slim abutments; by immunohistochemical quantification of T cells, B cells, macrophages, and PMNs.
Epithelial thickness and orientation of the collagen fibers | 3 months
  To compare the epithelial thickness and orientation of the collagen fibers of the peri-implant mucosa located around conventional and Slim abutments through a sample of peri-implant mucosa. One of the sections will be stained with HE, and we will use Image J image analysis software version 1.46 (U.S National Insitutes of Health, Bethesda, USA), calculating the mean of 25 thickness measurements for each of the samples. The other section will be stained with Masson-Goldner trichrome. With this staining, the light intensity will be increased for viewing the samples with a polarised light microscope. Collagen fibres aligned transverse to the direction of light propagation (parallel to the plane of section), will appear bright due to a change in the refraction of the existing light, whereas collagen fibres aligned along the axis of light propagation (perpendicular to the plane of section), will appear dark because no refraction occurs. Each sample will be observed at 5X, 10X, and 20W.
Vascular density of the peri-implant mucosa | 3 months
  To analyze and compare the vascular density of the peri-implant mucosa located around conventional esthetic abutments and the new Slim abutments through a sample of peri-implant mucosa by means of a section around the transepithelial abutment, with a circular biopsy scalpel of 6 mm diameter designed ad hoc, obtaining a sample of 1.5-2 mm.
Remnant soft tissue and/or microorganisms | 3 months
  To determine and compare the presence of remnant soft tissue and/or microorganisms on the surface of conventional esthetic abutments and the new Slim abutments we will use the SEM (Oxford Instruments INCA 300 EDX System, Abringdon, Oxfordshire, UK), and images will be captured using Semafore software (Semafore, JEOL, Tokyo, Japan).
Mesial and distal marginal bone loss | 36 months
  To clinically compare mesial and distal marginal bone loss using standardized digital periapical radiographs with parallel technique. Control at 12, 24 and 36 months.
Abutment stability | 3 months
  Basal and 3 months postimplantation measured by Implant Stability Quotient (ISQ).

CONTACTS AND LOCATIONS:
Overall Officials: Mario Pérez-Sayáns, PhD, Principal Investigator — University of Santiago de Compostela
Locations (1):
- Universidad de Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
We will anonymize and categorize the clinical data of the patients to share the information with the other researchers of the group
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Under request
Access Criteria: Under request